CLINICAL TRIAL: NCT05874063
Title: Thromboprophylaxis in Good and Intermediate Prognosis Advanced Germ Cell Tumors
Acronym: GIG-T
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-502426-41-00; CSET 2022/3510 (Other: Gustave Roussy ID)
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Germ Cell Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental for high-risk patients (Experimental): Thromboprophylaxis in addition of the standard chemotherapy
  Interventions: Drug: Thromboprophylaxis
- Control for high-risk patients (No Intervention): No thromboprophylaxis in addition of the standard chemotherapy
- Low-risk patients (No Intervention): No thromboprophylaxis in addition of the standard chemotherapy

INTERVENTIONS:
Drug: Thromboprophylaxis — Thromboprophylaxis in addition of the standard chemotherapy
  Arms: Experimental for high-risk patients

SUMMARY:
The goal of this clinical trial is to assess the efficacy of thromboprophylaxis in preventing venous thromboembolic events (VTE) in good and intermediate prognosis patients with metastatic germ cell cancer (GCT) undergoing first-line cisplatin-based chemotherapy with risk factors for developing a thromboembolic event .

The high-risk patients will be randomized between two treatments arm (receiving a thromboprophylaxis in the experimental arm, or no thromboprophylaxis in the control arm). The low-risk patients will be observed without any thromboprophylaxis. Patients will participate in the study for 14-17 weeks depending on the planned number of cycles of chemotherapy.

Researchers will compare an experimental arm with thromboprophylaxis and a control arm without thromboprophylaxis to detect an absolute decrease of 12% of the proportion of patients having experienced a VTE, from 21% (high risk patients, control arm) to 9% (high risk patients, experimental arm).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of good or intermediate prognosis of Germ Cell Tumor (according to the International Germ Cell Cancer Collaborative Group)
* Older than 18 years
* Suitable for first-line cisplatin-based chemotherapy
* No prior systemic cytotoxic therapy
* Additional criteria for patients who will be randomized (Venous Thromboembolic Event (VTE) high-risk patients): Lactate dehydrogenase higher than 1 Upper Normal Level and/or Body Surface Area higher than 1.9 and/or longer than 5 cm long axis retroperitoneal lymph nodes
* Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

* Brain metastasis
* History of VTE
* Concomitant use of anticoagulants or antiaggregants
* Renal impairment defined as creatinine clearance less than 50 ml/min using Cockcroft-Gault formula
* Hypersensitivity to enoxaparin sodium, heparin or its derivatives, including other low molecular weight heparins (LMWH) or to any of the excipients
* Any major surgery (i.e. open surgery lasting more than 45 minutes from opening to closure) within 4 weeks or planned during the study treatment period
* Severe uncontrolled high blood pressure (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg)
* Low baseline platelet count (< 100 X 10^9 /L) or history of heparin-induced thrombocytopenia
* Active clinically significant bleeding and conditions with a high risk of haemorrhage, including recent haemorrhagic stroke, gastrointestinal ulcer, presence of malignant neoplasm at high risk of bleeding, recent brain, spinal or ophthalmic surgery, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities
* Extensive metastatic disease at high risk of bleeding, e.g. prevalent choriocarcinoma
* Participation in another clinical study with an investigational product during the last 4 weeks, and while on study treatment without the approval from sponsor
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients undergoing a thromboembolic event | from randomization up to 6 weeks after D1 of the last cycle of chemotherapy or up to the residual masses surgery, whichever occurs first.
  (composite end point: symptomatic or asymptomatic (incidental finding) venous thrombosis or pulmonary embolism or unexplained death)

CONTACTS AND LOCATIONS:
Overall Officials: Karim FIZAZI, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (26):
- France (26):
  - ICO Paul Papin, Angers
  - CH de la Côte Basque, Bayonne
  - Institut Bergonié, Bordeaux
  - CHU de Brest, Brest
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital Tenon, Paris
  - CHU de Poitiers, Poitiers
  - Clinique La Croix du Sud, Quint-Fonsegrives
  - Institut Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - CHU de St Etienne, Saint-Etienne
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - HIA Bégin, Saint-Mandé
  - ICANS, Strasbourg
  - Hôpital Foch, Suresnes
  - Oncopole Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No